CLINICAL TRIAL: NCT04887909
Title: Prediction of Postoperative Visual Acuity in Cataract Patients Using a Macular Optical Coherence Tomography-based Deep Learning Method
Status: Not yet recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0496
Record Dates: First submitted 2021-05-13; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Data Collecting
Keywords: artificial intelligence; deep learning; cataract surgery; acuity vision; macular; optical coherence tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect the macular OCT images and preoperative and postoperative visual acuity of cataract patients who had been operated in the eye center of the Second Affiliated Hospital of Zhejiang University Medical College, and to train a model that can relatively accurately predict the postoperative visual acuity of patients by deep learing.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract patients, with or without macular disease, the impact of cataract on vision has affected the daily life of patients.

Exclusion Criteria:

* Glasses can obviously improve eyesight
* In addition to macular disease, combined with other eye diseases that seriously affect vision, resulting in no significant improvement in postoperative vision
* Complicated cataract surgery due to trauma and other reasons
* Combined with other eye diseases not suitable for intraocular lens implantation
* Patients with systemic diseases who cannot tolerate surgery

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cataract surgery was performed in ophthalmic hospital affiliated to Medical College of Zhejiang University
Sampling Method: Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2021-05-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Uncorrected distance visual acuity | 1 month postoperatively
  The UCVA was measured by the same optometrist at each visit
Best Corrected Visual Acuity | 1 month postoperatively
  The BCVA was measured by the same optometrist at each visit
Macular optical coherence tomography | 1 month postoperatively
  Macular oct was measured by the same doctor at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, China